CLINICAL TRIAL: NCT03563339
Title: Development and Pilot Test of Internet-delivered Postpartum Anxiety Prevention
Brief Title: Internet-delivered Postpartum Anxiety Prevention
Acronym: PPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Shari Steinman Haxel, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1710795361
Record Dates: First submitted 2018-05-29; First posted 2018-06-20 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Postpartum Disorder
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P-POD (Experimental): All participants will complete the prevention for postpartum onset distress (P-POD)
  Interventions: Behavioral: P-POD

INTERVENTIONS:
Behavioral: P-POD — . P-POD will include seven 30-minute online, educational, interactive modules that teach at-risk pregnant women skills derived from the gold standard, empirically supported cognitive-behavioral treatment for anxiety disorders and OCD. Additionally, P-POD will include three modules for fathers, to help them support their partners during the postpartum period. We will modify P-POD from an already existing in-person prevention program for postpartum OCD (developed by Co-Investigator Kiara Timpano). The m-health foundation of P-POD will be an already existing Internet-delivered treatment infrastructure (OurRelationship.com, developed by Co-Investigator Brian Doss).

SUMMARY:
Postpartum anxiety disorders are the most prevalent postpartum psychiatric conditions. Up to 16% of mothers experience postpartum anxiety or related disorders, such as OCD. With respect to the investigator's own community, this means that up to 3,313 women in West Virginia may struggle with postpartum anxiety or OCD. Left untreated, perinatal anxiety and OCD are associated with numerous adverse outcomes, such as maternal depression, preterm birth, impaired fetal development, low birthweight, difficulty breastfeeding, anxiety in children, and interference with parent-infant bonding. Critically, anxiety is a risk factor for cardiovascular disease and substance use disorders, both significant West Virginia health disparities. Thus, there is a critical need to develop effective and scalable prevention programs to address postpartum anxiety and OCD. The purpose of this proposed community-engaged study is to develop and test the feasibility, usability, and acceptability of an Internet-delivered postpartum anxiety and OCD prevention program, called "Preventing Postpartum Onset Distress", or P-POD.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 or older
* Pregnant with first child
* Married or living with a partner
* State Trait Anxiety Inventory-Trait Total ≥ 44 and/or Obsessive Beliefs Questionnaire-44 Total ≥ 139

Exclusion Criteria:

* past or current anxiety disorders
* past or current OCD
* past or current psychotic disorders
* past or current bipolar disorders
* past or current substance use disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 19 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory-Trait (STAI-Trait) | Change from Baseline to Week 10
  20-item self-report used to assess dispositional levels of anxiety. It is widely used, sensitive to treatment, has strong psychometric properties, and includes items that would be relevant to pregnant women. The STAI-Trait Total Score will be used before and after P-POD to assess change in prenatal trait anxiety. The STAI-Trait total score ranges from 20 to 80. Higher numbers represent more anxiety (worse outcome).
Obsessive Beliefs Questionnaire (OBQ-44) | Change from Baseline to Week 10
  44-item self-report scale used to measure dysfunctional beliefs associated with anxiety and OCD symptoms. The OBQ-44 has strong psychometric properties and has demonstrated sensitivity to treatment with pregnant women. In the proposed study, the OBQ-44 Total Score will be administered before and after P-POD to assess change in dysfunctional beliefs. The OBQ-44 total score ranges from 44 to 308. Higher numbers represent more dysfunctional OCD beliefs (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Life Sciences Building, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes